CLINICAL TRIAL: NCT01317641
Title: Safety and Pharmacokinetics of ODM-201 in Patients With Castrate Resistant Prostate Cancer: Open, Non-randomised, Uncontrolled, Multicentre, Multiple Dose Escalation Study With a Randomised Phase II Expansion Component
Brief Title: Safety and Pharmacokinetics Study of ODM-201 in Castrate Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Collaborators: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3104001
Record Dates: First submitted 2011-03-07; First posted 2011-03-17 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ODM-201 Phase I (Experimental)
  Interventions: Drug: ODM-201
- ODM-201 Phase II Dose 1 (Experimental)
  Interventions: Drug: ODM-201
- ODM-201 Phase II Dose 2 (Experimental)
  Interventions: Drug: ODM-201
- ODM-201 Phase II Dose 3 (Experimental)
  Interventions: Drug: ODM-201

INTERVENTIONS:
Drug: ODM-201 — ODM-201 administered orally daily

SUMMARY:
The purpose of this study is to evaluate safety, tolerability and pharmacokinetics of ODM-201 in patients with castrate resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Histologically confirmed adenocarcinoma of prostate
* Ongoing androgen deprivation therapy with a LHRH analogue or antagonist or bilateral orchiectomy
* Progressive metastatic disease
* Adequate bone marrow, hepatic, and renal function

Exclusion Criteria:

* Known metastases in the brain
* History of other malignancy within the previous 5 years
* Known gastrointestinal disease or procedure that affects the absorption
* Not able to swallow the study drug

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2011-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karim Fizazi, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (23):
- United States (8):
  - The Urology Center of Colorado, Wheat Ridge, Colorado
  - Eastern CT Hematology and Oncology Associates, Norwich, Connecticut
  - Urology Health Team PLLC, Ocala, Florida
  - Chesapeake Urology Research Associates, Baltimore, Maryland
  - Delaware Valley urology, LLC, Voorhees Township, New Jersey
  - Brooklyn Urology Research Group, Brooklyn, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
- Czechia (3):
  - Klinika onkologie a radioterapie LFUK a FN, Hradec Králové
  - Fakultni Nemonicnice Olomouc, Olomouc
  - Oddeleni Radiacni a Klinicke Onkologie Nemocnice Znojmo, Znojmo
- East-Tallinn Central Hospital, Talinn, Estonia
- Finland (5):
  - Helsinki University Central Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- France (2):
  - Saint Louis Hospital, Paris
  - Institut Gustave Roussy, Villejuif
- United Kingdom (4):
  - Queen Elizabeth Hospital, Birmingham
  - Velindre Cancer Centre, Cardiff
  - Christie Hospital, Manchester
  - Churchill Hospital, Oxford

REFERENCES:
- [Derived] Fizazi K, Massard C, Bono P, Jones R, Kataja V, James N, Garcia JA, Protheroe A, Tammela TL, Elliott T, Mattila L, Aspegren J, Vuorela A, Langmuir P, Mustonen M; ARADES study group. Activity and safety of ODM-201 in patients with progressive metastatic castration-resistant prostate cancer (ARADES): an open-label phase 1 dose-escalation and randomised phase 2 dose expansion trial. Lancet Oncol. 2014 Aug;15(9):975-85. doi: 10.1016/S1470-2045(14)70240-2. Epub 2014 Jun 25. PMID 24974051
- See also: PubMed link to the Lancet Oncology publication containing study results — http://www.ncbi.nlm.nih.gov/pubmed/24974051

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 23 hospitals in Europe and in the USA from Apr 5, 2011 to Mar 12, 2013
Pre-assignment Details: 136 participants participated in the study, including 24 enrolled in Phase 1 and 112 in Phase 2 randomly assigned to 200 mg, 400 mg or 1400 mg daily doses and stratified by previous chemotherapy and treatment with CYP17 inhibitor. Two participants assigned to treatment did not start ODM-201, and were therefore excluded from analyses populations.
Groups:
- Phase 1: ODM-201 200 mg/Day; Phase 1: ODM-201 400 mg/Day; Phase 1: ODM-201 600 mg/Day; Phase 1: ODM-201 1000 mg/Day; Phase 1: ODM-201 1400 mg/Day; Phase 1: ODM-201 1800 mg/Day: Dose escalation
- Phase 2: ODM-201 200mg/Day; Phase 2: ODM-201 400mg/Day; Phase 2: ODM-201 1400mg/Day: Chemotherapy-naïve and CYP17 inhibitor-naïve, Post-chemotherapy and CYP17 inhibitor-naïve, Post-CYP17 inhibitor
Period: Overall Study
Arm/Group | Phase 1: ODM-201 200 mg/Day | Phase 1: ODM-201 400 mg/Day | Phase 1: ODM-201 600 mg/Day | Phase 1: ODM-201 1000 mg/Day | Phase 1: ODM-201 1400 mg/Day | Phase 1: ODM-201 1800 mg/Day | Phase 2: ODM-201 200mg/Day | Phase 2: ODM-201 400mg/Day | Phase 2: ODM-201 1400mg/Day
Started | 4 | 7 | 3 | 4 | 3 | 3 | 38 | 38 | 36
Completed | 3 | 6 | 3 | 3 | 3 | 3 | 35 | 33 | 31
Not Completed | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 5 | 5
Not completed — Not treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Disease progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety
Groups:
- Phase 1, 200mg/Day ODM-201; Phase 1, 400mg/Day ODM-201; Phase 1, 600mg/Day ODM-201; Phase 1, 1000mg/Day ODM-201; Phase 1, 1400mg/Day ODM-201; Phase 1, 1800mg/Day ODM-201: Dose escalation. Participants received twice daily of oral ODM-201 continuously.
- Phase 2 (200mg/Day ODM-201); Phase 2 (400mg/Day ODM-201); Phase 2 (1400mg/Day ODM-201): Dose expansion. Participants received twice daily of 200 mg of oral ODM-201 continuously
- Total: Total of all reporting groups
Arm/Group | Phase 1, 200mg/Day ODM-201 | Phase 1, 400mg/Day ODM-201 | Phase 1, 600mg/Day ODM-201 | Phase 1, 1000mg/Day ODM-201 | Phase 1, 1400mg/Day ODM-201 | Phase 1, 1800mg/Day ODM-201 | Phase 2 (200mg/Day ODM-201) | Phase 2 (400mg/Day ODM-201) | Phase 2 (1400mg/Day ODM-201) | Total
Number analyzed (Participants) | 4 | 7 | 3 | 4 | 3 | 3 | 38 | 37 | 35 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (1.4) | 71.9 (8.5) | 65.3 (3.5) | 65.8 (11.2) | 67.7 (5.5) | 67.7 (3.2) | 68.3 (7.0) | 69.1 (7.4) | 71.3 (8.0) | 69.4 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 4 | 7 | 3 | 4 | 3 | 3 | 38 | 37 | 35 | 134

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants Who Experienced Dose Limiting Toxicity (DLT)
Description: A DLT was any Grade 3 or more toxicity (by National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE version 4.03]) excluding less than Grade 4 neutropenia or thrombocytopenia, hematological toxicity lasting less than 7 days, and nausea, vomiting, diarrhea controlled with antiemetic and/or anti-diarrheal treatment.
Time Frame: Up to 28 days for each cohort
Population: Safety population included all participants in Phase 1 who received any study drug.
Measure: Number; unit: events
Groups:
- Phase 1: ODM-201 200 mg/Day; Phase 1: ODM-201 400 mg/Day; Phase 1: ODM-201 600 mg/Day; Phase 1: ODM-201 1000 mg/Day; Phase 1: ODM-201 1400 mg/Day; Phase 1: ODM-201 1800 mg/Day: Participants received twice daily of oral ODM-201 continuously.
Arm/Group | Phase 1: ODM-201 200 mg/Day | Phase 1: ODM-201 400 mg/Day | Phase 1: ODM-201 600 mg/Day | Phase 1: ODM-201 1000 mg/Day | Phase 1: ODM-201 1400 mg/Day | Phase 1: ODM-201 1800 mg/Day
Number analyzed (Participants) | 4 | 7 | 3 | 4 | 3 | 3
events | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Phase 1: Number of Dose Limiting Toxicities Used to Determine the Maximum Tolerated Dose
Description: The MTD is defined as dose level at which 2 or more out of 6 participants experience a dose limiting toxicity (DLT)
Time Frame: Up to 28 days for each cohort
Population: Safety population included all participants in Phase 1 who received any study drug.
Measure: Number; unit: DLTs
Arm/Group | Phase 1: ODM-201 200 mg/Day | Phase 1: ODM-201 400 mg/Day | Phase 1: ODM-201 600 mg/Day | Phase 1: ODM-201 1000 mg/Day | Phase 1: ODM-201 1400 mg/Day | Phase 1: ODM-201 1800 mg/Day
Number analyzed (Participants) | 4 | 7 | 3 | 4 | 3 | 3
DLTs | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Phase 1 and 2: Participants With Decline of at Least 50% in Prostate-specific Antigen (PSA) in Chemotherapy-naïve and CYP17i-naïve Group
Description: Number of participants with greater than or equal to 50% decrease in serum PSA from baseline at 12 weeks in group of participants who were naïve to both chemotherapy and CYP17 inhibitor
Time Frame: 3 months
Population: Evaluable chemotherapy-naïve and CYP17i-naïve patients
Measure: Number; unit: participants
Groups:
- 200mg/Day ODM-201; 400mg/Day ODM-201; 1400mg/Day ODM-201: expanded dose level (phase 1 + phase 2)
- 600mg/Day ODM-201; 1000mg/Day ODM-201; 1800mg/Day ODM-201: phase 1
Arm/Group | 200mg/Day ODM-201 | 400mg/Day ODM-201 | 600mg/Day ODM-201 | 1000mg/Day ODM-201 | 1400mg/Day ODM-201 | 1800mg/Day ODM-201
Number analyzed (Participants) | 12 | 13 | 2 | 1 | 7 | 2
participants | 6 | 9 | 1 | 1 | 6 | 2

4. Secondary Outcome: Phase 1 and 2: Participants With Decline of at Least 50% in Prostate-specific Antigen (PSA) in Post-chemotherapy and CYP17i-naïve Group
Description: Number of participants with greater than or equal to 50% decrease in serum PSA from baseline at 12 weeks in group of participants previously treated with chemotherapy but not CYP17 inhibitor
Time Frame: 3 months
Population: Evaluable post-chemotherapy and CYP17i-naïve patients
Measure: Number; unit: participants
Arm/Group | 200mg/Day ODM-201 | 400mg/Day ODM-201 | 600mg/Day ODM-201 | 1000mg/Day ODM-201 | 1400mg/Day ODM-201 | 1800mg/Day ODM-201
Number analyzed (Participants) | 11 | 9 | 1 | 1 | 11 | 1
participants | 5 | 1 | 1 | 1 | 4 | 0

5. Secondary Outcome: Phase 1 and 2: Participants With Decline of at Least 50% in Prostate-specific Antigen (PSA) in Post-CYP17i Group
Description: Number of participants with greater than or equal to 50% decrease in serum PSA from baseline at 12 weeks in group of participants previously treated with CYP17 inhibitor
Time Frame: 3 months
Population: Evaluable post-CYP17 inhibitor patients
Measure: Number; unit: participants
Arm/Group | 200mg/Day ODM-201 | 400mg/Day ODM-201 | 1000mg/Day ODM-201 | 1400mg/Day ODM-201
Number analyzed (Participants) | 15 | 17 | 1 | 15
participants | 0 | 3 | 0 | 1

6. Secondary Outcome: Phase 1 and 2: Participants With RECIST Response in Soft Tissue in Chemotherapy-naïve and CYP17i-naïve Group
Description: Number of participants with overall complete response (CR), partial response (PR) or stable (SD) soft tissue disease according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) in chest, abdomen, and pelvic CT or MRI scans.
Time Frame: 3 months
Population: Evaluable Chemotherapy-naïve and CYP17i-naïve patients
Measure: Number; unit: participants
Arm/Group | 200mg/Day ODM-201 | 400mg/Day ODM-201 | 600mg/Day ODM-201 | 1400mg/Day ODM-201 | 1800mg/Day ODM-201
Number analyzed (Participants) | 9 | 9 | 2 | 2 | 2
participants
  RECIST response CR+PR | 1 | 4 | 0 | 1 | 0
  RECIST response CR+PR+SD | 9 | 6 | 2 | 2 | 2

7. Secondary Outcome: Phase 1 and 2: Participants With RECIST Response in Soft Tissue in Post-chemotherapy and CYP17i-naive Group
Description: as for outcome 6
Time Frame: 3 months
Population: Evaluable Post-chemotherapy and CYP17i-naïve patients
Measure: Number; unit: participants
Arm/Group | 200mg/Day ODM-201 | 400mg/Day ODM-201 | 1000mg/Day ODM-201 | 1400mg/Day ODM-201 | 1800mg/Day ODM-201
Number analyzed (Participants) | 8 | 7 | 1 | 5 | 1
participants
  RECIST response CR+PR | 1 | 0 | 0 | 1 | 0
  RECIST response CR+PR+SD | 5 | 3 | 0 | 4 | 1

8. Secondary Outcome: Phase 1 and 2: Participants With RECIST Responses in Soft Tissue in Post-CYP17i Group
Description: as for outcome 6
Time Frame: 3 months
Population: Evaluable Post-CYP17i patients
Measure: Number; unit: participants
Arm/Group | 200mg/Day ODM-201 | 400mg/Day ODM-201 | 1400mg/Day ODM-201
Number analyzed (Participants) | 13 | 12 | 9
participants
  RECIST response CR+PR | 0 | 2 | 0
  RECIST response CR+PR+SD | 5 | 9 | 6

9. Secondary Outcome: Phase 1 and 2: Participants With Stable Bone Disease in Chemotherapy-naïve and CYP17i-naïve Group
Description: Number of participants with stable bone disease (no change). Radiographic bone progression was defined by the appearance of two or more new lesions on bone scan
Time Frame: 3 months
Population: Evaluable chemotherapy-naïve and CYP17i-naïve patients with bone metastasis at baseline
Measure: Number; unit: participants
Arm/Group | 200mg/Day ODM-201 | 400mg/Day ODM-201 | 1000mg/Day ODM-201 | 1400mg/Day ODM-201 | 1800mg/Day ODM-201
Number analyzed (Participants) | 11 | 10 | 1 | 7 | 1
participants | 10 | 7 | 1 | 6 | 1

10. Secondary Outcome: Phase 1 and 2: Participants With Stable Bone Disease in Post-chemotherapy and CYP17i-naïve Group
Description: as for outcome 9
Time Frame: 3 months
Population: Evaluable Post-chemotherapy and CYP17i-naïve patients with bone metastasis at baseline
Measure: Number; unit: participants
Arm/Group | 200mg/Day ODM-201 | 400mg/Day ODM-201 | 600mg/Day ODM-201 | 1000mg/Day ODM-201 | 1400mg/Day ODM-201
Number analyzed (Participants) | 9 | 7 | 1 | 1 | 10
participants | 5 | 4 | 1 | 0 | 7

11. Secondary Outcome: Phase 1 and 2: Participants With Stable Bone Disease in Post-CYP17i Group
Description: as for outcome 9
Time Frame: 3 months
Population: Evaluable post-CYP17i patients with bone metastasis at baseline
Measure: Number; unit: participants
Arm/Group | 200mg/Day ODM-201 | 400mg/Day ODM-201 | 1000mg/Day ODM-201 | 1400mg/Day ODM-201
Number analyzed (Participants) | 11 | 15 | 1 | 11
participants | 5 | 9 | 1 | 6

12. Secondary Outcome: Phase 1: Area Under the Plasma-Concentration-time Curve (AUCt) of ODM-201 at Steady-state
Description: AUC(0-8h)
Time Frame: Day 8 predose 0 h and 0.5, 1, 1.5, 2, 4, 6 and 8 h postdose
Population: PK population (Day 8)
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- 200 mg/Day ODM-201; 400 mg/Day ODM-201; 600 mg/Day ODM-201; 1000 mg/Day ODM-201; 1400 mg/Day ODM-201; 1800 mg/Day ODM-201: Phase 1
Arm/Group | 200 mg/Day ODM-201 | 400 mg/Day ODM-201 | 600 mg/Day ODM-201 | 1000 mg/Day ODM-201 | 1400 mg/Day ODM-201 | 1800 mg/Day ODM-201
Number analyzed (Participants) | 3 | 7 | 3 | 3 | 3 | 3
h*ng/mL | 6387.27 (742.01) | 10973.66 (5939.78) | 14205.99 (2127.26) | 14817.39 (4190.48) | 31764.82 (8714.06) | 28884.44 (4900.60)

13. Secondary Outcome: Phase 1: Maximum Plasma Concentration (Cmax) of ODM-201 at Steady-state
Time Frame: Day 8 predose 0 h and 0.5, 1, 1.5, 2, 4, 6 and 8 h postdose
Population: PK population (Day 8)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 200 mg/Day ODM-201 | 400 mg/Day ODM-201 | 600 mg/Day ODM-201 | 1000 mg/Day ODM-201 | 1400 mg/Day ODM-201 | 1800 mg/Day ODM-201
Number analyzed (Participants) | 3 | 7 | 3 | 3 | 3 | 3
ng/mL | 1011.67 (168.84) | 1757.57 (858.72) | 2033.00 (277.59) | 2392.33 (406.63) | 4459.00 (1163.10) | 4235.00 (617.80)

14. Secondary Outcome: Phase 1: Time to Reach the Maximum Observed Concentration (Tmax) of ODM-201 at Day 1
Time Frame: 1 day
Population: PK population (Day 1)
Measure: Median (Standard Deviation); unit: h
Arm/Group | 200 mg/Day ODM-201 | 400 mg/Day ODM-201 | 600 mg/Day ODM-201 | 1000 mg/Day ODM-201 | 1400 mg/Day ODM-201 | 1800 mg/Day ODM-201
Number analyzed (Participants) | 4 | 7 | 3 | 4 | 3 | 3
h | 3.00 (1.63) | 3.00 (0.73) | 3.00 (0.92) | 5.08 (1.47) | 3.00 (1.15) | 5.00 (1.51)

15. Secondary Outcome: Phase 1: Area Under the Plasma-Concentration-time Curve (AUCt) of Major Metabolite ORM-15341 at Steady-state
Description: AUC(0-8h)
Time Frame: Day 8 predose 0 h and 0.5, 1, 1.5, 2, 4, 6 and 8 h postdose
Population: PK population (Day 8)
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 200 mg/Day ODM-201 | 400 mg/Day ODM-201 | 600 mg/Day ODM-201 | 1000 mg/Day ODM-201 | 1400 mg/Day ODM-201 | 1800 mg/Day ODM-201
Number analyzed (Participants) | 3 | 7 | 3 | 3 | 3 | 3
h*ng/mL | 11754.23 (5161.80) | 15501.56 (2755.85) | 24902.56 (12129.79) | 29980.83 (11658.75) | 63531.81 (15798.30) | 64435.97 (22930.30)

16. Secondary Outcome: Phase 1: Maximum Plasma Concentration (Cmax) of Major Metabolite ORM-15341 at Steady-state
Time Frame: Day 8 predose 0 h and 0.5, 1, 1.5, 2, 4, 6 and 8 h postdose
Population: PK population (Day 8)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 200 mg/Day ODM-201 | 400 mg/Day ODM-201 | 600 mg/Day ODM-201 | 1000 mg/Day ODM-201 | 1400 mg/Day ODM-201 | 1800 mg/Day ODM-201
Number analyzed (Participants) | 3 | 7 | 3 | 3 | 3 | 3
ng/mL | 1850.00 (654.83) | 2491.43 (328.86) | 3963.33 (1935.21) | 4643.33 (1340.01) | 9336.67 (2054.27) | 9406.67 (3165.38)

17. Secondary Outcome: Phase 1: Time to Reach the Maximum Observed Concentration (Tmax) of Major Metabolite ORM-15341 at Day 1
Time Frame: 1 day
Population: PK population (Day 1)
Measure: Median (Standard Deviation); unit: h
Arm/Group | 200 mg/Day ODM-201 | 400 mg/Day ODM-201 | 600 mg/Day ODM-201 | 1000 mg/Day ODM-201 | 1400 mg/Day ODM-201 | 1800 mg/Day ODM-201
Number analyzed (Participants) | 4 | 7 | 3 | 4 | 3 | 3
h | 3.00 (1.63) | 1.52 (1.33) | 3.00 (0.92) | 5.04 (2.05) | 3.00 (1.15) | 5.00 (0.55)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Phase 1 dose escalation and Phase 2 per dose
Groups:
- Phase 1, 200mg/Day ODM-201; Phase 1, 400mg/Day ODM-201; Phase 1, 600mg/Day ODM-201; Phase 1, 1000mg/Day ODM-201; Phase 1, 1400mg/Day ODM-201; Phase 1, 1800mg/Day ODM-201: Dose escalation
- Phase 2, 200mg/Day ODM-201; Phase 2, 400mg/Day ODM-201; Phase 2, 1400mg/Day ODM-201: Dose expansion
Arm/Group | Phase 1, 200mg/Day ODM-201 | Phase 1, 400mg/Day ODM-201 | Phase 1, 600mg/Day ODM-201 | Phase 1, 1000mg/Day ODM-201 | Phase 1, 1400mg/Day ODM-201 | Phase 1, 1800mg/Day ODM-201 | Phase 2, 200mg/Day ODM-201 | Phase 2, 400mg/Day ODM-201 | Phase 2, 1400mg/Day ODM-201
Serious Adverse Events (participants affected / at risk) | 0/4 | 2/7 | 0/3 | 1/4 | 1/3 | 0/3 | 2/38 | 3/37 | 4/35
Other Adverse Events (participants affected / at risk) | 4/4 | 5/7 | 2/3 | 4/4 | 3/3 | 2/3 | 33/38 | 35/37 | 27/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1, 200mg/Day ODM-201 (N=4) | Phase 1, 400mg/Day ODM-201 (N=7) | Phase 1, 600mg/Day ODM-201 (N=3) | Phase 1, 1000mg/Day ODM-201 (N=4) | Phase 1, 1400mg/Day ODM-201 (N=3) | Phase 1, 1800mg/Day ODM-201 (N=3) | Phase 2, 200mg/Day ODM-201 (N=38) | Phase 2, 400mg/Day ODM-201 (N=37) | Phase 2, 1400mg/Day ODM-201 (N=35)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1, 200mg/Day ODM-201 (N=4) | Phase 1, 400mg/Day ODM-201 (N=7) | Phase 1, 600mg/Day ODM-201 (N=3) | Phase 1, 1000mg/Day ODM-201 (N=4) | Phase 1, 1400mg/Day ODM-201 (N=3) | Phase 1, 1800mg/Day ODM-201 (N=3) | Phase 2, 200mg/Day ODM-201 (N=38) | Phase 2, 400mg/Day ODM-201 (N=37) | Phase 2, 1400mg/Day ODM-201 (N=35)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 5 | 6 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 1 | 0 | 0 | 2 | 0 | 4 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 4 | 4 | 3
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 7 | 8 | 5
Oedema peripheral (General disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 4
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 4
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 5
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 6 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 3
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 2
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 4 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Asthenia (General disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tinea cruris (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urine output increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other